CLINICAL TRIAL: NCT05658549
Title: Effect of N-Acetylcysteine on Neutrophil Lymphocyte Ratio And Length of Stay In COVID-19 Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, Head of Hospital Research Unit, Universitas Sebelas Maret
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAP02
Record Dates: First submitted 2022-11-26; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This research was an observational analytic cohort retrospective study in which the subjects were moderate degree COVID-19 inpatients in Sebelas Maret University Hospital divided into four groups. The control group K0 received standard therapy without NAC, while the treatment group, K1, received NAC injections of 1200mg/day, K2 NAC tablets 3x400mg/day, and K3 NAC tablets 3x200mg/day. Different tests using Way ANOVA and LSD or Kruskal-Wallis and Mann-Whitney.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study used N acetyl cysteine capsules and placebo, which were made similar in shape; researchers and patients did not know who was getting the drug or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- N-acetylcysteine injection 1200 mg (Experimental): N-acetylcysteine injection 1200 mg per day
  Interventions: Drug: N-acetyl cysteine
- N-acetylcysteine pill 1200 mg (Experimental): N-acetylcysteine pill 1200 mg orally per day
  Interventions: Drug: N-acetyl cysteine
- N-acetylcysteine pills 600 mg per day (Experimental): N-acetylcysteine pills 600 mg per day orally
  Interventions: Drug: N-acetyl cysteine
- placebo (Placebo Comparator): Capsule with shape and appearance similar to N-acetylcysteine
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine — N-acetyl cysteine dosage 600 mg and 1200 mg

SUMMARY:
This research is a study that compares the administration of N-acetylcysteine at various doses with the outcomes of COVID-19 patients, namely the neutrophil-to-lymphocyte ratio and length of stay.

DETAILED DESCRIPTION:
This research was an observational analytic cohort retrospective study in which the subjects were moderate degree COVID-19 inpatients in Sebelas Maret University Hospital divided into four groups. The control group K0 received standard therapy without NAC, while the treatment group K1 received NAC injections of 1200mg/day, K2 NAC tablets 3x400mg/day, and K3 NAC tablets 3x200mg/day. Different tests using Way ANOVA and LSD or Kruskal-Wallis and Mann-Whitney.

ELIGIBILITY:
Inclusion Criteria:

* moderate or severe grade confirmed COVID-19 (patients with symptoms and radiological examination showing pneumonia with or without signs of severe pneumonia: SpO2<90%, respiratory rate>30x/min, and severe respiratory distress) who were admitted to UNS Hospital and age 18-60 years old

Exclusion Criteria:

* patients who died during the treatment period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Neutrophil to lymphocyte ratio | Change of Neutrophil to lymphocyte ratio at 7 day
  Neutrophil to lymphocyte ratio
Length of stay | From date of randomization until the date of return from hospital
  Length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Sebelas Maret Hospital, Sukoharjo, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No